CLINICAL TRIAL: NCT04283643
Title: Noninvasive Brain Stimulation for Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21311
Record Dates: First submitted 2020-02-03; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pain, Acute; Pain, Chronic; Pain, Experimental
Keywords: Transcranial Magnetic Stimulation; Focused Ultrasound; Noninvasive Neuromodulation
MeSH Terms: conditions — Acute Pain; Chronic Pain; Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Within subjects design of real and control stimulation, pain measures and behavioral assessments may be compared between healthy subjects and pain groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Human Subjects (Experimental): Healthy human subjects will complete study procedures in the research lab at UVA. They will complete pain-related behavioral questionnaires and undergo experimental pain testing for temperature and laser stimuli for real and control conditions of brain stimulation.
  Interventions: Other: Transcranial Focused Ultrasound; Other: Transcranial Magnetic Stimulation
- Acute Pain Patients (Experimental): Acute Pain Patients will complete study procedures in the hospital or clinic at UVA. They will complete pain-related behavioral questionnaires and undergo experimental pain testing for temperature and laser stimuli for real and control conditions of brain stimulation, as well as rate their ongoing pain.
  Interventions: Other: Transcranial Focused Ultrasound; Other: Transcranial Magnetic Stimulation
- Chronic Pain Patients (Experimental): Chronic Pain Patients will complete study procedures in the hospital or clinic at UVA. They will complete pain-related behavioral questionnaires and undergo experimental pain testing for temperature and laser stimuli for real and control conditions of brain stimulation, as well as rate their ongoing pain.
  Interventions: Other: Transcranial Focused Ultrasound; Other: Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Transcranial Focused Ultrasound — Non-invasive brain stimulation technique
Other: Transcranial Magnetic Stimulation — Non-invasive brain stimulation technique

SUMMARY:
Non-invasive brain stimulation techniques, transcranial magnetic stimulation (TMS) and transcranial focused ultrasound (FUS), is be applied to healthy human subjects, acute pain patients, and chronic pain patients to investigate their uses for pain relief.

DETAILED DESCRIPTION:
The research team will be using non-invasive brain stimulation techniques, transcranial magnetic stimulation (TMS) and transcranial focused ultrasound (FUS) to investigate their uses for pain relief in humans: healthy human subjects, acute pain patients, and chronic pain patients. Magnetic Resonance Imaging (MRI) and electroencephalogram (EEG) recordings will be collected to achieve the following objectives:

Objective 1 aims to determine the effects of noninvasive brain stimulation on the pain-related brain activities during pain processing. We hypothesize that noninvasive brain stimulation approaches will increase or decrease cortical activity upon processing painful input.

Objective 2 aims to determine the effects of noninvasive brain stimulation on pain intensity and/or pain-related behavioral assessments. We hypothesize that noninvasive brain stimulation will influence pain-intensity and/or pain-related behavioral assessments.

Objective 3 aims to investigate the correlation between brain activity and pain relief after noninvasive brain stimulation. We hypothesize that noninvasive brain stimulation will suppress cortical activity in pain-related brain areas, reduce pain intensity, and/or improve pain-related behavioral assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 80 years of age.
* Chronic and Acute pain patients: must have an MRI (for ultrasound targeting)

Exclusion Criteria:

* Direct report to the study team member
* History of brain surgery
* History of seizure
* Pregnant
* Have alcohol consumption exceeding 50 drinks/month
* Have history of opioid abuse (all subjects), or any recent opioid use (healthy controls)
* Have implant like pacemaker and aneurysm clip
* Current of psychiatric disease such as anxiety or depression, which is not optimally treated
* Current infection
* Current wound on the skin of upper and lower extremities
* Chronic pain patients: current chronic pain is not optimal controlled by pain medications (i.e. Pain VAS >5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | immediately after brain stimulation (same day, approximately 5-10 minutes after baseline) as compared to baseline
  Participants will rate their pain (experimental, acute, chronic) on a 1-10 scale
Numeric Pain Rating Scale | immediately after experimental pain measure (up to 15 minutes after baseline) as compared to baseline
  Participants will rate their pain (experimental, acute, chronic) on a 1-10 scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided